CLINICAL TRIAL: NCT02400372
Title: The Effect of Anti-bacterial Honey Dressing on the Healing of Split Thickness Skin Graft Donor Site
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0079-14
Record Dates: First submitted 2015-02-10; First posted 2015-03-27 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Disorder of Skin Donor Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- research group (Experimental): Medihoney Dressing
  Interventions: Device: medihoney dressing
- control group (No Intervention): Paraffin gauze with saline Dressing
- 3. Comparison group (No Intervention): Polymem dressing

INTERVENTIONS:
Device: medihoney dressing — to evaluate the effect of medihoney dressing on the healing of split thickness skin graft donor site
  Arms: research group

SUMMARY:
The study, "Evaluation of the effect of antibacterial medical honey dressing for healing of implants donor area", is a Phase 4 Study, Prospective, A randomized trial, 3 arms (treatment groups) trial, Open-label, non-controlled, non-randomized, Aims To test the effectiveness of antibacterial medical honey dressing in the therapy of donor area of implants. In our Research Will participate in 135 new patients over the age of 18, with a wound in the donor area of hip implants, Hospitalized in the Plastic Surgery Unit of the "Haemek" Medical Center. Appropriate patients, who will agree to sign and sign a consent form, be assigned randomly to one of three treatment groups:

1. The research group: Medihoney antibacterial wound dressing.
2. The control group: Paraffin gauze with saline- The basic treatment in the donor site, accepted the literature.
3. Comparison group: Polymem dressing - Common treatment in the donor site in the Plastic Surgery Unit of the "Haemek" Medical Center.

Participants in the three study groups will be performed, each visit, Medical monitoring and examination by a team of medical indices of Plastic Surgery Unit, as is customary. The treatment will be performed, twice a week until recovery and the complete closure of the wound.

DETAILED DESCRIPTION:
Study protocol The aim of this study is to evaluate "The effect of anti-bacterial honey dressing on the healing of split thickness skin graft donor site".

Protocol Abstract. The use of skin grafts for wound closure is considered one of the common methods in the field of plastic surgery. Healing of the donor area is secondary, gradual and is a serious problem, Associated with a high percentage of wound infections, Delay in healing, Scars, Pain unpleasant odor and other problems. As of today, there is no ideal treatment to cure the donor area of implants, due to lack of high-quality comparative studies. The use of honey to treat wounds known for centuries in different cultures. Honey has anti-inflammatory and anti-bacterial effect, Debridement ability, and Pain relief. Honey has almost no side effects. Effectiveness of honey in wound healing has been tested in many clinical trials, but most of them and some methodological problems of low quality. Therefore, it is difficult to conclude that the existing information handling guidelines and recommending further clinical research.

The study, "Evaluation of the effect of antibacterial medical honey dressing for healing of implants donor area", is a Phase 4 Study, Prospective, A randomized trial, 3 arms (treatment groups) trial, Open-label, non-controlled, non-randomized, Aims To test the effectiveness of antibacterial medical honey dressing in the therapy of donor area of implants. In our Research Will participate in 135 new patients over the age of 18, with a wound in the donor area of hip implants, Hospitalized in the Plastic Surgery Unit of the "Haemek" Medical Center. Appropriate patients, who will agree to sign and sign a consent form, be assigned randomly to one of three treatment groups:

1. The research group: Medihoney antibacterial wound dressing.
2. The control group: Paraffin gauze with saline- The basic treatment in the donor site, accepted the literature.
3. Comparison group: Polymem dressing - Common treatment in the donor site in the Plastic Surgery Unit of the "Haemek" Medical Center.

Participants in the three study groups will be performed, each visit, Medical monitoring and examination by a team of medical indices of Plastic Surgery Unit, as is customary. The treatment will be performed, twice a week until recovery and the complete closure of the wound.

Research Goals Primary goal Examining the effect of Medihoney antibacterial wound dressing honey on the duration of the donor site area healing, until full recovery and wound closure.

Secondary objectives

1. To Evaluatee the effect of Medihoney antibacterial wound dressing on pain intensity donor site.
2. . To Evaluatee the effect of Medihoney antibacterial wound dressing on the frequency of infections in donor site.

Tertiary goal

1. To evaluate the effect of Medihoney antibacterial wound dressing on the unpleasant odor in the donor site.
2. 2. To evaluate the effect of Medihoney antibacterial wound dressing on patient satisfaction from treatment in donor site.

Research Hypothesis Medihoney antibacterial wound dressing will find significantly statistical more effective in comparison with Paraffin gauze with saline dressing and compared with Polymem dressing, In terms of duration of a treatment, Intensity of pain and the prevalence of infection in the donor site.

Treatment regimen First group Immediately after harvesting the skin, the donor site will be covered with a thin layer of Medihoney Antibacterial Wound Gel and Xtrasorb Super Absorbent Dressing will used as secondary dressing. After 24 hours, the dressing will be replaced by Medihoney HCS dressing.

Medihoney HCS dressing will be replace twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a wound on the hip - the implant donor area
* Wound size up to 100 sm²

Exclusion Criteria:

* Known sensitivity of the patient to honey
* Pregnant women
* Patients under 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Examining the effect of Medihoney antibacterial wound dressing honey on the duration of the donor site area healing, until full recovery and wound closure | 25 days
  The Outcome will be assessed by Medical examination and Laboratory Testing

SECONDARY OUTCOMES:
To Evaluatee the effect of Medihoney antibacterial wound dressing on the frequency of infections in donor site. | 25 days
  The Outcome will be assessed by Medical examination and Laboratory Testing
To Evaluatee the effect of Medihoney antibacterial wound dressing on pain intensity donor site. | 25 days
  The Outcome will be assessed by Medical examination and Questionnaire
To evaluate the effect of Medihoney antibacterial wound dressing on the unpleasant odor in the donor site. | 25 days
  The Outcome will be assessed by Medical examination and Questionnaire
To evaluate the effect of Medihoney antibacterial wound dressing on patient satisfaction from treatment in donor site. | 25 days
  The Outcome will be assessed by Medical examination and Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Shufani, MD, Principal Investigator — HaEmek Medical Center, Afula
Locations (1):
- HaEmekMC, Afula, Israel